CLINICAL TRIAL: NCT06543147
Title: The Effect of Education About Breast Cancer and Breast Self- Examination on Breast Cancer Fear and Health Beliefs: Randomized Controlled Trial
Brief Title: Effect of Education on Breast Cancer Fear and Health Beliefs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Collaborators: Ordu University Scientific Research Projects Coordination Department (Unknown)
Responsible Party: Principal Investigator, Nermin Kayar, RN, Msc., Lecturer, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Nermin KAYAR; 2018/B-1838 (Other Grant/Funding Number: Ordu University Scientific Research Projects Coordination Department)
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Women's Health; Health Education
Keywords: Breast self examination; health belief model; breast cancer; breast cancer fear
MeSH Terms: conditions — Health Education; Breast Self-Examination; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Administering a pre-test to the participants in the experimental and control groups. After the pre-test, the participants in the experimental group were given breast cancer and breast self-examination training, brochure distribution, and reminders of breast self-examination by phone for six months. They administered a post-test to the participants in the experimental and control groups six months later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): There are 79 female participants in this group. After the pre-test, participants in the experimental group were given breast cancer and breast self-examination training. After the training, they were reminded to do breast self-examination by phone for six months. The post-test was administered six months later.
  Interventions: Other: breast cancer and breast self- examination education
- Control Group (No Intervention): There are 80 female participants in this group. A pre-test was applied to the participants in the control group. The participants in the experimental group were given an intervention for six months, while the participants in the control group were not. A post-test was applied after six months. Based on the principle of sufficient and accurate care, women in the control group were given training about breast cancer and BSE in groups of 7-9 people after posttest data were collected and given brochures at the end of training

INTERVENTIONS:
Other: breast cancer and breast self- examination education — The experimental group were given education about breast cancer and BSE. Slide presentations used during training provided information about breast anatomy and physiology, breast cancer symptoms and risk factors, early diagnosis methods for breast cancer and breast cancer screening programs, and barriers to breast cancer screening programs were discussed. In addition to slide presentations about breast cancer and BSE, women were also given BSE training on a breast examination mannequin and given brochures after training. The training lasted 40-50 minutes. After women in the experimental group were given training, they were called by telephone once per month until 6 months and reminded about doing BSE.
  Arms: experimental group

SUMMARY:
The study was conducted to determine the effect of breast cancer and breast self-examination (BSE) education on breast cancer fear and health beliefs. The main questions it aims to answer are:

H1: Breast cancer and BSE training given to women will affect the health beliefs of women.

H2: Breast cancer and BSE training given to women will affect the fear of breast cancer among women.

H3: Breast cancer and BSE training given to women will affect the information and behaviour in relation to breast cancer screening among women.

Researchers divided participants into experimental and control groups to examine the effects of breast cancer and breast self-examination education on breast cancer fear and health beliefs. The experimental group received education about breast cancer and breast self-examination and was reminded to perform breast self-examination by phone for six months.

DETAILED DESCRIPTION:
Before beginning the research, women were informed about the aim, duration, and procedures during the research and they were included in the research after written consent was obtained from women accepting participation. Then pre-test data were collected. The collection of data in the research began on 16 October 2017.

In the first stage of the research, pre-test data were collected using the questionnaire form, Champion Health Belief Model Scale, Champion Breast Cancer Fear Scale, and face-to-face interview method, and women were asked to fill out the forms themselves. After the pre-test data were collected, the women were divided into experimental and control groups using a single-blind randomized method.

In the second stage of the research, women in the experimental group were given education about breast cancer and BSE. Slide presentations used during training provided information about breast anatomy and physiology, breast cancer symptoms and risk factors, early diagnosis methods for breast cancer and breast cancer screening programs, and barriers to breast cancer screening programs were discussed. In addition to slide presentations about breast cancer and BSE, women were also given BSE training on a breast examination mannequin and given brochures after training. The training lasted 40-50 minutes. Training was given in groups of 7-9 people and was completed from 2 April 2018 to 30 April 2018. After women in the experimental group were given training, they were called by telephone once per month until 6 months and reminded about doing BSE.

In the final stage of the research, a post-test was applied to women in the experiment and control groups six months after the first training. The posttest applied the questionnaire, CHBMS, and CBCFS for a second time. Attempts were made to determine the effect of the training and counseling on breast cancer health beliefs and fear of breast cancer.

Based on the principle of sufficient and accurate care, women in the control group were given training about breast cancer and BSE in groups of 7-9 people after posttest data were collected and given brochures at the end of training

ELIGIBILITY:
Inclusion Criteria:

* Being over 20 years old
* not having a history of breast cancer
* not being in the lactation process
* not having a communication barrier
* volunteering to participate in the study

Exclusion Criteria:

* having a history of breast cancer
* having a communication barrier
* being in the lactation process
* not volunteering to participate in the study

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — based on self-representation
Enrollment: 160 (Actual)
Dates: Start 2018-03-17 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Champion Health Belief Model Scale | Six mounth
  The CHBMS consists of 6 subscales and 42 items; susceptibility perception of the perceived individual risks of catching breast cancer (3 items), seriousness perception about the perceived degree of individual threat from breast cancer (7 items), benefits perception expressing advantages related to BSE (4 items), barriers perception about perceived obstacles related to BSE (11 items), confidence expressing perceived individual competence in the ability to identify an abnormal breast mass during BSE (10 items) and health motivation subscale (7 items). Each subscale is evaluated separately and total points including the whole scale are not calculated. Women receiving low points for the barrier subscale and high points from the other subscales show positive attitudes and beliefs related to breast cancer and BSE
Champion Breast Cancer Fear Scale | Six mounth
  Items on the scale investigate emotions like fear, upset, tension, irritation, restlessness, and worry and situations like depression or increased heart rate when breast cancer is considered. The scale contains 8 items and has a five-point Likert response. Responses to the scale are "definitely disagree" 1 point, "disagree" 2 points, "undecided" 3 points, "agree" 4 points and "completely disagree" 5 points. The lowest points that can be obtained from the scale is 8 with the highest points of 40. High points show high levels of fear about breast cancer. For definition of fear levels to breast cancer low levels of fear are 8-15 points, moderate levels of fear are 16-23 points and high levels of fear are 24-40 points.

CONTACTS AND LOCATIONS:
Overall Officials: nermin kayar, Principal Investigator — nerminkayar@klu.edu.tr
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Clinical data are not publicly available due to privacy laws. Questions regarding data can be directed to the corresponding author.

REFERENCES:
- [Background] Karayurt O, Dramali A. Adaptation of Champion's Health Belief Model Scale for Turkish women and evaluation of the selected variables associated with breast self-examination. Cancer Nurs. 2007 Jan-Feb;30(1):69-77. doi: 10.1097/00002820-200701000-00013. PMID 17235224
- [Result] Champion VL, Skinner CS, Menon U, Rawl S, Giesler RB, Monahan P, Daggy J. A breast cancer fear scale: psychometric development. J Health Psychol. 2004 Nov;9(6):753-62. doi: 10.1177/1359105304045383. PMID 15367754